CLINICAL TRIAL: NCT04668885
Title: Lower Doses of CPX-351 as a Novel Approach for the Treatment of Older Patients With Relapsed or Refractory Acute Myeloid Leukemia and Myelodysplastic Syndromes
Brief Title: CPX-351 as a Novel Approach for the Treatment of Older Patients With AML and MDS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE1920
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Refractory Acute Myeloid Leukemia; Relapsed Acute Myelomonocytic Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Myelodysplastic Syndromes | interventions — CPX-351

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Primary refractory/relapsed AML (Experimental): Lower dose CPX-351 in participants with primary refractory/relapsed AML. Participants will receive an induction and maintenance phase of CPX-351
  Interventions: Drug: CPX-351
- MDS after HMA failure (Experimental): Lower dose CPX-351 in participants with MDS after HMA failure. Participants will receive an induction and maintenance phase of CPX-351
  Interventions: Drug: CPX-351

INTERVENTIONS:
Drug: CPX-351 — Induction phase: CPX-351 15 mg/m^2 on days 1 and 3 of each 28-day cycle for up to a total of 6 cycles in the absence of unacceptable toxicity
  Maintenance phase: CPX-351 7.5 mg/m^2 on days 1 and 3 for two cycles alternating with 15 mg/m^2 for one cycle. Participants may receive up to 12 cycles of maintenance phase in the absence of unacceptable toxicity.

SUMMARY:
The purpose of this study is to evaluate how effective lower doses of CPX-351 are in older participants with relapsed/refractory acute myeloid leukemia (AML) who are not eligible to receive intensive chemotherapy and in participants with myelodysplastic syndromes (MDS) after Hypomethylating Agents (HMA) failure.

DETAILED DESCRIPTION:
Currently, elderly patients with AML and high risk MDS, who are ineligible to receive induction chemotherapy and fail HMA +/- combination, have very poor outcomes and there is no FDA-approved therapy outside of some targeted therapies which can only be applied to a small patient population. CPX-351 is an investigational (experimental) drug that works by combining two anti-cancer drugs cytarabine and daunorubicin. CPX-351 is experimental because it is only FDA approved for the treatment of adults with two types of AML: newly diagnosed therapy-related AML or AML with myelodysplasia-related changes.

This is an open label clinical trial of lower doses of CPX-351 in relapsed/primary refractory older AML and MDS patients ineligible to receive intensive chemotherapy. The first arm is for particpants with primary refractory/relapsed AML and the second arm is for higher risk MDS participants after HMA failure.

ELIGIBILITY:
Inclusion Criteria:

* Primary refractory or relapsed AML (defined by 2016 World Health Organization [WHO] criteria) patients who are not suitable for or not willing to receive intensive chemotherapy as evaluated by the treating physician. Primary refractory disease is defined as:

  * Failure to achieve a CR, CRi, or mLFS (defined as <5% Bone Marrow (BM) blasts) after receiving 1 or 2 cycles of remission induction chemotherapy.
  * Failure to achieve a CR, CRi, or MLFS (defined as <5% BM blasts) after receiving 4 cycles of non-intensive chemotherapy or whose disease progressed at any time point during the treatment.
* Participants with MDS (according to 2016 WHO criteria) who did not respond to treatment with azacitidine, decitabine, or combination of HMA with another drug or lost their response to initial therapy with HMA.
* Eastern Cooperative Oncology Group (ECOG) performance status <=2
* Adequate hepatic (serum total bilirubin < 1.5 x ULN, Serum glutamic pyruvic transaminase (SGPT) and/or serum glutamate oxaloacetate transaminase (SGOT) <2.5 x ULN) and renal function (creatinine < 1.5mg/dL).
* Participants must be willing and able to review, understand, and provide written consent before starting therapy.

Exclusion Criteria:

* Active signs or symptoms of central nervous system (CNS) involvement by malignancy (lumbar puncture [LP] not required).
* Prior 7+3 remission induction chemotherapy for MDS or AML
* More than 2 lines of prior non-intensive therapy.
* New York Heart Association (NYHA) class III or IV heart disease, active ischemia or any other uncontrolled cardiac condition such as angina pectoris, clinically significant cardiac arrhythmia on rhythm control strategy or on pacemaker, uncontrolled hypertension (blood pressure > 160 systolic and > 110 diastolic not responsive to antihypertensive medication)
* Acute myocardial infarction in the previous 12 weeks (from the start of treatment).
* Any serious medical condition, laboratory abnormality, or psychiatric illness that, in the view of the treating physician, would place the participant at an unacceptable risk if he or she were to participate in the study or would prevent that person from giving informed consent.
* Any active malignancy (unrelated, non-hematological malignancy) diagnosed within the past 6 months of starting the study drug (other than curatively treated carcinoma-in-situ of the cervix or non-melanoma skin cancer).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CPX-351.
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known history of HIV or active hepatitis B or C.
* No major surgery within 2 weeks prior to study enrollment.
* Pregnant or breast feeding
* Male and female participants who are fertile who do not agree to use an effective barrier methods of birth control (i.e. abstinence) to avoid pregnancy while receiving study treatment and for 30 days after last dose of study treatment. Non-childbearing is defined as > 1 year postmenopausal or surgically sterilized.
* Acute promyelocytic leukemia (APL)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) per 2003 International Working Group (IWG) criteria | At 6 months
  ORR = complete response (CR) + CR with incomplete blood count recovery (CRi) + partial remission (PR) as defined by 2003 IWG criteria for AML patients, and ORR = CR + PR + hematologic improvement (HI) and as defined per 2006 IWG criteria for MDS patients
Overall response rate (ORR) per 2003 IWG criteria | At 1 year
  ORR = complete response (CR) + CR with incomplete blood count recovery (CRi) + partial remission (PR) as defined by 2003 IWG criteria for AML patients, and ORR = CR + PR + hematologic improvement (HI) and as defined per 2006 IWG criteria for MDS patients
Overall response rate (ORR) per 2003 IWG criteria | At 1.5 years
  ORR = complete response (CR) + CR with incomplete blood count recovery (CRi) + partial remission (PR) as defined by 2003 IWG criteria for AML patients, and ORR = CR + PR + hematologic improvement (HI) and as defined per 2006 IWG criteria for MDS patients
Overall response rate (ORR) per 2003 IWG criteria | At 2 years
  ORR = complete response (CR) + CR with incomplete blood count recovery (CRi) + partial remission (PR) as defined by 2003 IWG criteria for AML patients, and ORR = CR + PR + hematologic improvement (HI) and as defined per 2006 IWG criteria for MDS patients
Overall response rate (ORR) per 2003 IWG criteria | At 2.5 years
  ORR = complete response (CR) + CR with incomplete blood count recovery (CRi) + partial remission (PR) as defined by 2003 IWG criteria for AML patients, and ORR = CR + PR + hematologic improvement (HI) and as defined per 2006 IWG criteria for MDS patients
Overall response rate (ORR) per 2003 IWG criteria | At 3 years
  ORR = complete response (CR) + CR with incomplete blood count recovery (CRi) + partial remission (PR) as defined by 2003 IWG criteria for AML patients, and ORR = CR + PR + hematologic improvement (HI) and as defined per 2006 IWG criteria for MDS patients
Overall response rate (ORR) per 2003 IWG criteria | At 3.5 years
  ORR = complete response (CR) + CR with incomplete blood count recovery (CRi) + partial remission (PR) as defined by 2003 IWG criteria for AML patients, and ORR = CR + PR + hematologic improvement (HI) and as defined per 2006 IWG criteria for MDS patients
Overall response rate (ORR) per 2003 IWG criteria | At 4 years
  ORR = complete response (CR) + CR with incomplete blood count recovery (CRi) + partial remission (PR) as defined by 2003 IWG criteria for AML patients, and ORR = CR + PR + hematologic improvement (HI) and as defined per 2006 IWG criteria for MDS patients
Overall response rate (ORR) per 2003 IWG criteria | At 4.5 years
  ORR = complete response (CR) + CR with incomplete blood count recovery (CRi) + partial remission (PR) as defined by 2003 IWG criteria for AML patients, and ORR = CR + PR + hematologic improvement (HI) and as defined per 2006 IWG criteria for MDS patients
Overall response rate (ORR) per 2003 IWG criteria | At 5 years
  ORR = complete response (CR) + CR with incomplete blood count recovery (CRi) + partial remission (PR) as defined by 2003 IWG criteria for AML patients, and ORR = CR + PR + hematologic improvement (HI) and as defined per 2006 IWG criteria for MDS patients

SECONDARY OUTCOMES:
Time to response (TTR) | At 6 months
  TTR is measured from start of treatment to the date of achieving a response. Wilcoxon rank test will be used for comparison of continuous variables.
Time to response (TTR) | At 1 year
  TTR is measured from start of treatment to the date of achieving a response. Wilcoxon rank test will be used for comparison of continuous variables.
Time to response (TTR) | At 1.5 years
  TTR is measured from start of treatment to the date of achieving a response. Wilcoxon rank test will be used for comparison of continuous variables.
Time to response (TTR) | At 2 years
  TTR is measured from start of treatment to the date of achieving a response. Wilcoxon rank test will be used for comparison of continuous variables.
Time to response (TTR) | At 2.5 years
  TTR is measured from start of treatment to the date of achieving a response. Wilcoxon rank test will be used for comparison of continuous variables.
Time to response (TTR) | At 3 years
  TTR is measured from start of treatment to the date of achieving a response. Wilcoxon rank test will be used for comparison of continuous variables.
Time to response (TTR) | At 3.5 years
  TTR is measured from start of treatment to the date of achieving a response. Wilcoxon rank test will be used for comparison of continuous variables.
Time to response (TTR) | At 4 years
  TTR is measured from start of treatment to the date of achieving a response. Wilcoxon rank test will be used for comparison of continuous variables.
Time to response (TTR) | At 4.5 years
  TTR is measured from start of treatment to the date of achieving a response. Wilcoxon rank test will be used for comparison of continuous variables.
Time to response (TTR) | At 5 years
  TTR is measured from start of treatment to the date of achieving a response. Wilcoxon rank test will be used for comparison of continuous variables.
Duration of response (DOR) | At 6 months
  DOR measured from the time of achieving a response to time of disease progression. Wilcoxon rank test will be used for comparison of continuous variables.
Duration of response (DOR) | At 1 year
  DOR measured from the time of achieving a response to time of disease progression. Wilcoxon rank test will be used for comparison of continuous variables.
Duration of response (DOR) | At 1.5 years
  DOR measured from the time of achieving a response to time of disease progression. Wilcoxon rank test will be used for comparison of continuous variables.
Duration of response (DOR) | At 2 years
  DOR measured from the time of achieving a response to time of disease progression. Wilcoxon rank test will be used for comparison of continuous variables.
Duration of response (DOR) | At 2.5 years
  DOR measured from the time of achieving a response to time of disease progression. Wilcoxon rank test will be used for comparison of continuous variables.
Duration of response (DOR) | At 3 years
  DOR measured from the time of achieving a response to time of disease progression. Wilcoxon rank test will be used for comparison of continuous variables.
Duration of response (DOR) | At 3.5 years
  DOR measured from the time of achieving a response to time of disease progression. Wilcoxon rank test will be used for comparison of continuous variables.
Duration of response (DOR) | At 4 years
  DOR measured from the time of achieving a response to time of disease progression. Wilcoxon rank test will be used for comparison of continuous variables.
Duration of response (DOR) | At 4.5 years
  DOR measured from the time of achieving a response to time of disease progression. Wilcoxon rank test will be used for comparison of continuous variables.
Duration of response (DOR) | At 5 years
  DOR measured from the time of achieving a response to time of disease progression. Wilcoxon rank test will be used for comparison of continuous variables.
Event-free survival (EFS) | At 6 months
  EFS measured from date of first dose to the date of treatment failure, relapse, or death from any cause. Wilcoxon rank test will be used for comparison of continuous variables
Event-free survival (EFS) | At 1 year
  EFS measured from date of first dose to the date of treatment failure, relapse, or death from any cause. Wilcoxon rank test will be used for comparison of continuous variables
Event-free survival (EFS) | At 1.5 years
  EFS measured from date of first dose to the date of treatment failure, relapse, or death from any cause. Wilcoxon rank test will be used for comparison of continuous variables
Event-free survival (EFS) | At 2 years
  EFS measured from date of first dose to the date of treatment failure, relapse, or death from any cause. Wilcoxon rank test will be used for comparison of continuous variables
Event-free survival (EFS) | At 2.5 years
  EFS measured from date of first dose to the date of treatment failure, relapse, or death from any cause. Wilcoxon rank test will be used for comparison of continuous variables
Event-free survival (EFS) | At 3 years
  EFS measured from date of first dose to the date of treatment failure, relapse, or death from any cause. Wilcoxon rank test will be used for comparison of continuous variables
Event-free survival (EFS) | At 3.5 years
  EFS measured from date of first dose to the date of treatment failure, relapse, or death from any cause. Wilcoxon rank test will be used for comparison of continuous variables
Event-free survival (EFS) | At 4 years
  EFS measured from date of first dose to the date of treatment failure, relapse, or death from any cause. Wilcoxon rank test will be used for comparison of continuous variables
Event-free survival (EFS) | At 4.5 years
  EFS measured from date of first dose to the date of treatment failure, relapse, or death from any cause. Wilcoxon rank test will be used for comparison of continuous variables
Event-free survival (EFS) | At 5 years
  EFS measured from date of first dose to the date of treatment failure, relapse, or death from any cause. Wilcoxon rank test will be used for comparison of continuous variables
Overall Survival (OS) | At 6 months
  OS measured from start of treatment to death or last follow up. OS function will be estimated using the Kaplan-Meier method
Overall Survival (OS) | At 1 year
  OS measured from start of treatment to death or last follow up. OS function will be estimated using the Kaplan-Meier method
Overall Survival (OS) | At 1.5 years
  OS measured from start of treatment to death or last follow up. OS function will be estimated using the Kaplan-Meier method
Overall Survival (OS) | At 2 years
  OS measured from start of treatment to death or last follow up. OS function will be estimated using the Kaplan-Meier method
Overall Survival (OS) | At 2.5 years
  OS measured from start of treatment to death or last follow up. OS function will be estimated using the Kaplan-Meier method
Overall Survival (OS) | At 3 years
  OS measured from start of treatment to death or last follow up. OS function will be estimated using the Kaplan-Meier method
Overall Survival (OS) | At 3.5 years
  OS measured from start of treatment to death or last follow up. OS function will be estimated using the Kaplan-Meier method
Overall Survival (OS) | At 4 years
  OS measured from start of treatment to death or last follow up. OS function will be estimated using the Kaplan-Meier method
Overall Survival (OS) | At 4.5 years
  OS measured from start of treatment to death or last follow up. OS function will be estimated using the Kaplan-Meier method
Overall Survival (OS) | At 5 years
  OS measured from start of treatment to death or last follow up. OS function will be estimated using the Kaplan-Meier method

CONTACTS AND LOCATIONS:
Overall Officials: Sudipto Mukherjee, MD, PhD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual patient data in order to protect the confidentiality of the participants who enroll on this study